CLINICAL TRIAL: NCT01901770
Title: The Ohio State University Center for Population Health and Health Disparities Community Awareness, Resources and Education (CARE II): Project 4 The PARENT (Parents in Appalachia Receive Education Needed for Teens) Project
Brief Title: The Parents in Appalachia Receive Education Needed for Teen Project
Acronym: PARENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-11115; NCI-2013-01164 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-07-13; First posted 2013-07-17 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Human Papilloma Virus Infection
Keywords: HPV; Ohio Appalachia; HPV vaccine; No evidence of disease
MeSH Terms: conditions — Papillomavirus Infections | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I-HPV vaccine education (Experimental): The educational intervention is that parents and providers receive materials about HPV by mail including HPV/ cervical cancer videos and brochures, fact sheets, HPV/cervical cancer resource lists. Clinics receive posters, brochures, tabletop/reminder cards, resource lists, newsletters, and "invitation to be vaccinated" letters for parents.
  Interventions: Other: educational intervention
- Arm II- Flu vaccine education (Active Comparator): The educational intervention is that parents and providers receive materials about Flu by mail including Flu brochures, fact sheets, Flu resource lists. Clinics receive posters and brochures.
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — Receive HPV vaccination educational materials
  Other Names: intervention, educational
  Arms: Arm I-HPV vaccine education
Other: educational intervention — Receive influenza vaccination educational materials
  Other Names: intervention, educational
  Arms: Arm II- Flu vaccine education

SUMMARY:
This clinical trial studies an educational intervention for parents and providers in increasing human papillomavirus (HPV) vaccination rates in younger girls in Ohio Appalachia. Educational interventions may be effective in increasing the number of participants whose daughters receive HPV vaccination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Implement a multi-level HPV vaccine educational intervention directed at 3 levels within participating 12 Ohio Appalachia counties that includes information about cervical cancer, cervical cancer screening, HPV, the HPV vaccine, communication skills training to improve parent-health care provider conversations about the HPV vaccine, and organizational level components.

II. Evaluate the effectiveness of the multi-level HPV vaccine educational intervention in a group randomized controlled trial in 12 Ohio Appalachia counties.

OUTLINE: Participants are randomized to 1 of 2 arms.

Arm I: Parents and health care providers receive educational materials about HPV vaccination by mail or in-person review with project staff including a culturally tailored HPV and cervical cancer educational video and brochures, a question and answer (Q & A) fact sheet, and a HPV and cervical cancer resource list. Clinics receive waiting and exam room posters and brochures, tabletop cards, reminder cards to mail to participants, an information resource list, newsletter, vaccine tracking system, and "invitation to be vaccinated" letter to mail to parents.

Arm II: Parents and health care providers receive educational materials about influenza vaccination by mail or in-person review with project staff.

After completion of study, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* LEVEL 1: Parents
* Be able to speak, read, and write English
* Has a daughter who receives care from or lives in one of 12 Ohio Appalachia counties
* Be a parent or a guardian of a young girl (age 9 to 17 years) who has not received the HPV vaccine (if a parent has more than one daughter, they will be asked questions about their eldest daughter)
* Not have a child who has received the HPV vaccine

LEVEL 2: Health care providers

* Practicing in a participating public health department or provider office in Ohio Appalachia
* Personnel involved in the vaccine process (determined by individual health departments or clinic)
* Able to speak, read, and write English

Exclusion Criteria:

LEVEL 1: Parents

* Not able to speak, read, and write English
* Does not have a daughter who receives care from or lives in one of 12 Ohio Appalachia counties
* Not the parent or a guardian of a young girl (age 9 to 17 years) who has not received the HPV vaccine (if a parent has more than one daughter, they will be asked questions about their eldest daughter)
* Has a child who has received the HPV vaccine

LEVEL 2: Health care providers

* Does not practicing in a participating public health department or provider office in Ohio Appalachia
* Personnel that is not involved in the vaccine process (determined by individual health departments or clinic)
* Not able to speak, read, and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2012-01; Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of daughters of participating parents who received their first HPV vaccination | Within 3 months of viewing educational material
  A logistic random effects model will be used. A t-test of the coefficient for intervention status will be used to determine if there is a difference in the expected proportion of vaccinated patients across treatment arms.

SECONDARY OUTCOMES:
Proportion of daughters of participants in the intervention arm who received a second and third dose of the HPV vaccine | Up to 6 months
  Separate logistic random effects models will be fit for each vaccination and t-tests of the fixed intervention effect will be used to compare treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Electra Paskett, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu